CLINICAL TRIAL: NCT01189799
Title: Motivational Therapy for Substance Users With Depression
Acronym: Aftercare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Suzette Glasner-Edwards, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1K23DA020085 (NIH); 1K23DA020085 (NIH)
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Depression; Substance Dependence
Keywords: Co-occurring Disorders; Depression; Substance Dependence; Motivational Therapy; Aftercare; Cognitive Behavioral Therapy
MeSH Terms: conditions — Depression; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Therapy Aftercare (Experimental): Twelve, 60 minute weekly structured manualized therapy sessions.
  Interventions: Behavioral: Motivational therapy
- Dual Recovery Anonymous/Tx as usual (Active Comparator): Aftercare Treatment as Usual,which is twelve 60 minute weekly sessions of peer led 12-step Dual Recovery Anonymous group.
  Interventions: Behavioral: Dual Recovery Anonymous/Tx as usual

INTERVENTIONS:
Behavioral: Motivational therapy — Twelve, 60 minute weekly structured manualized therapy sessions.
  Arms: Motivational Therapy Aftercare
Behavioral: Dual Recovery Anonymous/Tx as usual — Twelve 60 minute weekly sessions of peer led 12-step Dual Recovery Anonymous group.
  Arms: Dual Recovery Anonymous/Tx as usual

SUMMARY:
The primary objective of the study is to test the incremental efficacy and outcomes of an aftercare program of Cognitive Behavioral Therapy combined with motivational therapy (CBT-MT) relative to treatment as usual (TAU) in improving depression, substance use, and healthcare outcomes in a population with drug dependence and comorbid major depressive disorder (MDD). The investigators expect that among drug-dependent patients with comorbid MDD, CBT-MT will yield better clinical outcomes relative to TAU in reducing depressive symptoms and substance use and improving healthcare outcomes during treatment.

Secondary Objectives:

1. Test efficacy and outcomes of CBT-MT and TAU
2. Evaluate the differential effect of CBT-MT versus TAU on HIV-risk behavior of participants,
3. To evaluate the impact of cognitive functioning on treatment retention and outcomes, and
4. To explore additional psychosocial, demographic, and diagnostic factors (e.g., age, gender, education level, motivation for change, social support) that may be associated with treatment outcome and retention in this high need population.

DETAILED DESCRIPTION:
This study will include approximately 80 participants randomized to either 12 weeks of motivational therapy or treatment as usual. Both treatments will meet once weekly for 60 minutes. Participants will be recruited from the Adult Partial Hospitalization program at University of California, Los Angeles. During the active treatment phase, participants will attend clinic weekly for collection of data and urine specimens.

1. For those randomly assigned to CBT-MT, they will meet with a therapist in a group format for 60-minute sessions once weekly.

   a. Each CBT-MT session will begin with 20 minutes of motivational therapy (MT), followed by 40 minutes of CBT content.
2. Those randomly assigned to TAU, they will attend a weekly 60-minute Dual Recovery Anonymous self-help group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or over
2. DSM-IV diagnosis of Substance Dependence (cannabis, stimulant, opioid, or prescription drug) or DSM-IV diagnosis of Alcohol Dependence and abuse of cannabis, stimulant, opioid, or prescription drug
3. Diagnostic and Statistical Manual -IV diagnosis of lifetime Major Depressive Disorder (MDD)
4. BDI-II score of 13 or greater

Exclusion Criteria:

1. Presence of life threatening or unstable medical illness
2. Lack of proficiency in English
3. Current homelessness (unless residing in a recovery home for which contact information can be provided)
4. Psychiatric symptoms warranting safety concerns or inpatient treatment, including acute suicide risk
5. Present diagnosis of Bipolar Disorder, Schizophrenia, or Schizoaffective Disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in Substance Use | weekly during active phase and through study completion, up to 6 months
  * Participants will provide a sample for a urine drug screen (UDS).
  * Participants will also self report substance use.
Change in Depression symptoms | weekly during intervention and through study completion, up to 6 months
  -Participants will complete the Beck's Depression Inventory (BDI) to measure changes in depression symptoms over time.
Change in Healthcare utilization | weekly and at follow up, up to 6 months
  -Participants will self report use of ancillary treatment and healthcare services including ER visits and hospitalizations.

SECONDARY OUTCOMES:
Efficacy and outcomes of CBT-MT and TAU | Baseline, end of treatment, and at follow up, up to 6 months
  - Participants will complete the Addiction Severity Index to assess change in psychosocial functioning between baseline, end of treatment and follow up.
HIV-risk behavior of participants | Baseline, end of treatment and follow up, up to 6 months
  -Participants will complete the Risk Behavior Assessment (RBA) to measure effect of CBT-MT versus TAU on changes in HIV risk behaviors.
Cognitive functioning | Baseline and end of treatment at 3 months post treatment
  -Participants will complete the MicroCog and Wisconsin Card Sort Test impact of cognitive functioning on treatment retention and outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Glasner, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Integrated Substance Abuse Programs, Los Angeles, California, United States